CLINICAL TRIAL: NCT07068594
Title: The Effect of Virtual Reality Application on Pain, Anxiety, and Vital Parameters During the First Dressing Change After Open Heart Surgery
Brief Title: The Application of Virtual Reality Goggles During the First Wound Dressing After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Almira Gurcan, RN, MSc - Specialist Nurse in Surgical Nursing, Department of Surgical Diseases Nursing, Adnan Menderes University, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OHSFP2025-01; NoSecondaryID01 (Other: NoSecondaryID01)
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Pain Management; Wound Care; Heart Surgery; Heart Surgery Via Sternotomy; Dressing
Keywords: virtual reality; pain; anxiety; heart surgery; wound dressing; vital signs; nursing; intensive care unit nursing; surgical nursing
MeSH Terms: conditions — Agnosia; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Glasses During the First Dressing Change Usage (Experimental): In this group, virtual reality glasses were used during the procedure for individuals who would have their first dressing changed on the first postoperative day after open heart surgery.
  Interventions: Device: Virtual Reality Goggles
- Standard Dressing Procedure without VR (No Intervention): A standard dressing change procedure was performed on this group.

INTERVENTIONS:
Device: Virtual Reality Goggles — A device consisting of glasses placed on the head of patients in the intervention group and earphones attached to the glasses
  Arms: Virtual Reality Glasses During the First Dressing Change Usage

SUMMARY:
The aim of this study is to examine the effect of virtual reality glasses, a non-pharmacological method used in pain and anxiety management in nursing practices, on the pain, anxiety, and vital parameters perceived by patients undergoing their first dressing change after open heart surgery. Additionally, the study aims to obtain information about the safety of the virtual reality application. The primary questions this study seeks to answer are as follows:

Does the virtual reality headset application reduce the pain participants feel during the procedure?

Does the application reduce participants' anxiety levels during the procedure?

Does the virtual reality application have a positive effect on vital signs (pulse, blood pressure, etc.)?

Do participants experience any side effects or medical problems during this application?

Researchers will compare the group that received virtual reality glasses during the first dressing change after open-heart surgery with the standard care (control group) to evaluate the effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who verbally or in writing agree to participate in the study,
* Are over 18 years of age,
* Have not been diagnosed with any psychiatric disorder and are not using psychiatric medication,
* Have no visual, auditory, or perceptual impairments,
* Are undergoing their first wound dressing change following open-heart surgery,

Exclusion Criteria:

* Patients who are unconscious,
* Individuals who have undergone two or more wound dressing changes after open-heart surgery,
* Patients who report pain due to any other condition,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Immediately before the dressing procedure and 10 minutes after the procedure
  Pain intensity will be assessed using the Visual Analog Scale (VAS). It is a 10 cm scale ranging from 0 (no pain) to 10 (worst possible pain). Measurements were taken before the dressing procedure and 10 minutes after the procedure.

SECONDARY OUTCOMES:
Anxiety level | Immediately before the dressing procedure and 10 minutes after the procedure
  Anxiety will be measured using the State-Trait Anxiety Inventory (STAI). The inventory consist of 20 items rated on a 4 point Likert scale ranging from 1 (not at all), to 4 (very much so). The state anxiety subscale will be pre and post intervention to evaluate changes in situational anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydin Adnan Menderes University - Institute of Health Sciences, Aydin, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes